CLINICAL TRIAL: NCT01628627
Title: Long Term, Double Blind, Randomized, Placebo Controlled Multi-center Study of FRE.M.S.- Frequency Modulated Neural Stimulation Lorenz Therapy™ in Symptomatic Diabetic Neuropathy
Brief Title: Frequency Modulated Neural Stimulation (FREMS) in Symptomatic Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lorenz Biotech S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EuropeanFREMS
Record Dates: First submitted 2012-06-23; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FREMS (Experimental): Frequency Modulated Neural Stimulation (FREMS)
  Interventions: Device: Frequency Modulated Neural Stimulation (FREMS) (Aptiva)
- Control (Sham Comparator)
  Interventions: Device: sham treatment (Aptiva)

INTERVENTIONS:
Device: Frequency Modulated Neural Stimulation (FREMS) (Aptiva) — FREMS consisted of sequences of biphasic (negative and positive), asymmetric and electrically balanced pulses, composed of: 1) an active phase of high negative voltage spike (variable, max -300 V) and extra short duration (variable, 10-100 μsec, mostly ~40 μsec); followed by: 2) a recharging phase of low voltage and long duration (0.9 - 999 msec); pulse frequency was variable, ranging 1 to 1,000 Hz, mainly in the low range 1-50 Hz. Three cycles of 10 consecutive (one a day for 5 days/week) applications to both lower limbs were delivered.
  Other Names: Aptiva device (Lorenz Biotech, Medolla, Italy)
  Arms: FREMS
Device: sham treatment (Aptiva) — The sham treatment consisted of no electrical pulses delivered by the same device used to deliver the FREMS treatment and with the same treatment procedure and schedule.
  Other Names: Aptiva device (Lorenz Biotech, Medolla, Italy)
  Arms: Control

SUMMARY:
Aim of this study is to evaluate safety and efficacy of transcutaneous frequency modulated electromagnetic neural stimulation (FREMS) to treat symptomatic peripheral neuropathy in patients with diabetes mellitus.

DETAILED DESCRIPTION:
Diabetic neuropathy is a common and potentially disabling complication of patients with type 1 or type 2 diabetes due to the damage of peripheral nerves caused by chronic hyperglycemia. The most common clinical signs and symptoms of diabetic neuropathy include numbness, diminished sensation and painful symptoms, such as burning, pins and needles, intolerable pain and hyperaesthesia of the lower extremities.

Different classes of drugs, such as analgesics, antidepressants and anti-epileptics are variably efficacious in pain relief, but are unfortunately unable to revert the natural history of the disease.

A wide range of electrotherapies have been proposed for the non-pharmacological treatment of diabetic neuropathy. The rationale of using electric or magnetic stimulation is the potential enhancement of microcirculation and endoneural blood flow, possibly counteracting the nerve ischemic damage, together with other yet poorly understood mechanisms, such as masking pain by interfering with pain gate control.

A number of studies have reported the efficacy of different electrotherapies, such as transcutaneous electrical nerve stimulation (TENS), pulsed-dose electrical stimulation, peripheral nerve, nerve root, spinal cord, deep brain and epidural motor cortex stimulations, pulsed (electro-)magnetic fields and static magnetic fields, high-frequency external muscle stimulation, high-tone external muscle stimulation and external muscle stimulation. However, of all these electrotherapies, only TENS is currently recommended as a treatment for painful diabetic neuropathy by the American Academy of Neurology.

Recently, a novel transcutaneous frequency-modulated electromagnetic neural stimulation (also named as Frequency Rhythmic Electrical Modulation System, FREMS), has been developed. FREMS consists of a sequence of modulated electrical stimuli that varies automatically in terms of pulse frequency, duration and voltage amplitude. FREMS was tested in a pilot randomized, cross-over study, and reduced diabetic neuropathy pain and ameliorated the sensory tactile and vibration perception threshold and motor nerve conduction velocity compared to a sham treatment.

The aim of this study was to test the efficacy and safety of FREMS in a multicentre, randomized, double-blind, placebo-controlled study enrolling a large population with symptomatic diabetic polyneuropathy, with repeated treatment sessions and a post-treatment follow-up of adequate length.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes
* Diabetes duration of > 1 year
* Age: 18 to 75 years
* Symptomatic neuropathy
* Abnormal amplitude, latency or conduction velocity in at least one motor nerve (Tibial or Peroneal) or in the Sural Nerve
* A measurable Sural Nerve conduction velocity
* Stable glycemic control in the last 3 months, HbA1C < 11%
* MDNS score > 7
* Stable dose of analgesic medications, if any, in the month prior enrollment

Exclusion Criteria:

* Previous treatment with TENS or other electrotherapy
* Motor or Sensitive nerve conduction velocity < 30 non recordable/evocable
* Unstable glycemic control during last 3 months
* Pregnancy
* Implanted pacemaker or defibrillator or neurostimulator
* Cancer diagnosed in the last 5 years
* Psychological or psychiatric disorders that in the Investigator's opinion may interfere with patient's compliance to study procedures
* Active foot ulcer and/or major lower limb amputation
* Diabetic mononeuropathy
* Severe peripheral artery disease (Leriche Fontaine scale grade 3 and 4)
* Ankle-brachial index (ABI) < 0.7
* Uremic neuropathy or end-stage renal disease
* Toxic neuropathies
* Severe hepatic disease
* Alcohol consumption ≥ 40 g/day or 30 units/week

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in Nerve Conduction Velocity of the Deep Peroneal, Tibial, or Sural Nerve | baseline and 51 weeks
  Change in Nerve Conduction Velocity of the Deep Peroneal , Tibial, or Sural Nerve at 51 weeks (i.e., after three cycles of FREMS treatment) versus baseline

SECONDARY OUTCOMES:
Change in Vibration Perception Threshold | baseline and 51 weeks
  Change in Vibration Perception Threshold at 51 weeks (i.e., after three cycles of FREMS treatment) versus baseline
Change in Cold Sensory Threshold | baseline and 51 weeks
  Change in Cold Sensory Threshold at 51 weeks (i.e., after three cycles of FREMS treatment) versus baseline
Change in Warm Sensory Threshold | baseline and 51 weeks
  Change in Warm Sensory Threshold at 51 weeks (i.e., after three cycles of FREMS treatment) versus baseline
Change in Day Pain Intensity (Visual Analogue Scale) | baseline and week 3
  Change in Pain Intensity (assessed using Visual Analogue Scale) during day time with the first cycle of FREMS
Change in Day Pain Intensity (Visual Analogue Scale) | week 17 and week 20
  Change in Pain Intensity (assessed using Visual Analogue Scale) during day time with the second cycle of FREMS
Change in Day Pain Intensity (Visual Analogue Scale) | week 34 and week 37
  Change in Pain Intensity (assessed using Visual Analogue Scale) during day time with the third cycle of FREMS
Change in Night Pain Intensity (Visual Analogue Scale) | baseline and week 3
  Change in Pain Intensity (assessed using Visual Analogue Scale) during night time with the first cycle of FREMS
Change in Night Pain Intensity (Visual Analogue Scale) | week 17 and week 20
  Change in Pain Intensity (assessed using Visual Analogue Scale) during night time with the second cycle of FREMS
Change in Night Pain Intensity (Visual Analogue Scale) | week 34 and week 37
  Change in Pain Intensity (assessed using Visual Analogue Scale) during night time with the third cycle of FREMS
Change in the Michigan Diabetic Neuropathy Score (MDNS) | baseline and 51 weeks
  Change in the Michigan Diabetic Neuropathy Score (MDNS) at 51 weeks (i.e. after three FREMS cycles) versus baseline
Change in the dose and type of analgesic medications | baseline and 51 weeks
  Change in the dose and type of analgesic medications at week 51 (i.e. after three FREMS cycles) versus baseline
Number of patients with treatment-related adverse events | baseline and 51 weeks
  Change in the dose and type of analgesic medications at week 51 (i.e. after three FREMS cycles) versus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, MD, Principal Investigator — San Raffaele Hospital & Scientific Institute
Locations (6):
- Paris-Nord University, Bondy, Ile Del France, France
- Heinrich Heine University, Düsseldorf, Germany
- Italy (4):
  - San Raffaele Hospital & Scientific Institute, Milan, MI
  - University of Padua, Padua, PD
  - University of Perugia, Perugia, PG
  - Tor Vergata University, Rome, RM

REFERENCES:
- [Background] Conti M, Peretti E, Cazzetta G, Galimberti G, Vermigli C, Pola R, Scionti L, Bosi E. Frequency-modulated electromagnetic neural stimulation enhances cutaneous microvascular flow in patients with diabetic neuropathy. J Diabetes Complications. 2009 Jan-Feb;23(1):46-8. doi: 10.1016/j.jdiacomp.2008.02.004. Epub 2008 Apr 10. PMID 18403219
- [Background] Bosi E, Conti M, Vermigli C, Cazzetta G, Peretti E, Cordoni MC, Galimberti G, Scionti L. Effectiveness of frequency-modulated electromagnetic neural stimulation in the treatment of painful diabetic neuropathy. Diabetologia. 2005 May;48(5):817-23. doi: 10.1007/s00125-005-1734-2. Epub 2005 Apr 15. PMID 15834546
- [Derived] Bosi E, Bax G, Scionti L, Spallone V, Tesfaye S, Valensi P, Ziegler D; FREMS European Trial Study Group. Frequency-modulated electromagnetic neural stimulation (FREMS) as a treatment for symptomatic diabetic neuropathy: results from a double-blind, randomised, multicentre, long-term, placebo-controlled clinical trial. Diabetologia. 2013 Mar;56(3):467-75. doi: 10.1007/s00125-012-2795-7. Epub 2012 Dec 13. PMID 23238789